CLINICAL TRIAL: NCT06227325
Title: Prospective, Single Center, Phase II Study of Disitamab Vedotin（RC48) Combined With Sintilimab Plus XELOX for Perioperative Treatment of Locally Advanced Gastric Cancer With HER2 Overexpression
Brief Title: Disitamab Vedotin Combined With Sintilimab and XELOX Perioperative Treatment for Resectable Gastric Caner With HER2 Overexpression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCVDTYPEC067
Record Dates: First submitted 2024-01-11; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-09

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; XELOX

STUDY DESIGN:
Intervention Model Description: RC48+PD-1+chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Neoadjuvant therapy:RC48 combined with Sintilimab and XELOX repeat every 2 weeks or every 3 weeks for a total of 3 cycles Adjuvant therapy: RC48 combined with Sintilimab and XELOX repeat every 2 weeks or every 3 weeks for a total of 5 cycles
  Interventions: Drug: RC48 combined with Sintilimab and XELOX

INTERVENTIONS:
Drug: RC48 combined with Sintilimab and XELOX — RC48: 2.5 mg/kg, iv, d1, repeat every 2 weeks; Sintilimab: 200mg, iv, d1, repeat every 3 weeks; XELOX: Oxaliplatin 130mg/m2, iv, d1；Capecitabine1000 mg po, bid, d1-14, repeat every 3 weeks
  Other Names: Disitamab vedotin combined with Sintilimab and XELOX

SUMMARY:
The aim of this study is to observe the efficacy, safety, postoperative pathological response rate and survival benefit of RC48 combined withSintilimab and chemotherapy in perioperative therapy of locally advanced resectable gastric and gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects volunteered to join the study, could complete the signing of the informed consent form, and had good compliance;
2. Aged at least 18-75 years, male or female;
3. Gastric cancer or adenocarcinoma of gastroesophageal junction confirmed by histology and/or cytology is diagnosed as cT3-4aN1-3M0 according to AJCC version 8, and cTNM is diagnosed as cT3-4aN1-3M0 according to endoscopic ultrasonography or enhanced CT/MRI scanning (combined with ultrasonic gastroscopy and diagnostic laparoscopic exploration if necessary), and the researcher evaluates that the lesion is resectable;
4. Have not received systematic treatment for current diseases in the past, including surgical treatment, anti-tumor radiochemotherapy/immunotherapy, etc;
5. Patients who agree to receive radical surgical treatment and have no surgical contraindication as judged by the surgeon.
6. IHC(immuno-histochemistry) results confirmed HER2 expression (defined as IHC 2+and 3+);
7. ECOG (Eastern Cooperative Oncology Group) score 0-1;
8. Expected life ≥ 6 months;
9. The main organs function well and meet the standards:
10. The fertile subjects must use appropriate methods of contraception during the study period and within 120 days after the end of the study. The serum pregnancy test was negative within 7 days before the study was included, and they must be non lactating subjects.

Exclusion Criteria:

1. Malignant diseases other than gastric cancer diagnosed within 5 years prior to initial administration;
2. Known endoscopic signs of active bleeding;
3. The subject is currently participating in an interventional clinical study, or has received other investigational drugs or used investigational devices within 4 weeks prior to initial dosing;
4. Previous treatment with anti-HER2, anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs targeting another stimulus or synergistic inhibition of T cell receptors;
5. Received systemic systemic treatment with Chinese patent drugs with anti-tumor indications or immunomodulatory drugs (including thymosin, interferon, interleukin, except for local use to control pleural fluid) within 2 weeks before the first administration;
6. An active autoimmune disease requiring systemic treatment (e.g. with disease-modifying drugs, glucocorticoids, or immunosuppressants) has occurred within 2 years prior to first administration. Replacement therapies (such as thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy;
7. Was receiving systemic glucocorticoid therapy (excluding topical glucocorticoids by nasal spray, inhalation, or other route) or any other form of immunosuppressive therapy within 7 days prior to the study's initial administration;
8. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
9. Known allergy to the drugs used in this study;
10. Has not fully recovered from toxicity and/or complications caused by any intervention before starting treatment (i.e., ≤ grade 1 or baseline, excluding weakness or hair loss);
11. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);
12. Untreated active hepatitis B (defined as HBsAg positive and HBV(hepatitis B virus)-DNA copy number detected greater than the upper limit of normal value in the laboratory of the study center);
13. Active HCV-infected subjects (HCV antibody positive and HCV-RNA levels above the lower limit of detection);
14. Received live vaccine within 30 days prior to the first dose (cycle 1, day 1);
15. Pregnant or lactating women;
16. The presence of any serious or uncontrolled systemic disease;
17. Evidence of medical history or disease that might interfere with the test results, prevent participants from fully participating in the study, abnormal treatment or laboratory test values, or other conditions that the investigator considers unsuitable for enrollment The Investigator considers other potential risks unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) rate | Up to approximately 12 weeks
  The percentage of patients with no residual cells at the primary cancer site and N(-) per histological evaluation.

SECONDARY OUTCOMES:
R0 resection rate | Up to approximately 12 weeks
  The percentage of patients who have no residual cancer cells (gross or microscopically) at the resection margins.
Disease free survival (DFS) | From randomization to the date of recurrence or death (up to approximately 4 years).
  DFS is defined as the time from postoperative baseline imaging evaluation to disease recurrence or death in subjects who are disease-free after surgery.
Major pathological response (MPR) rate | Up to approximately 12 weeks
Clinical downgrading rate | Up to approximately 12 weeks
Overall survival (OS) | From the randomization to the date of death (up to approximately 4 years).
  OS is defined as the time from the first dose to all-cause death.
Percentage of Participants who experience one or more adverse events (AEs). | Up to approximately 2 years
  The incidence and grade of adverse events (including SAE) will be determined per NCI-CTCAE 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Liu, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China